CLINICAL TRIAL: NCT00912717
Title: The Pancreatic Adenocarcinoma Gene Environment Risk Study -A Prospective Cohort Study of Patients at Risk or Having Pancreatic Disease
Brief Title: Pancreatic Adenocarcinoma Gene Environment Risk Study
Acronym: PAGER
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Randall Brand, M.D., University of Pittsburgh
Other Study IDs: STUDY19070256
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pancreatic Cancer: individuals who have been diagnosed with pancreatic cancer
- Unaffected: individuals who have not been diagnosed with pancreatic cancer

SUMMARY:
After informed consent, participants will be asked to complete a medical/family history questionnaire and provide a blood sample. Some participants may also be asked to provide a urine sample. Individuals undergoing procedures that require collection of biological samples for clinical purposes may have these samples saved for research purposes. Participants will also be asked for their permission for study investigators to access medical records and/or recontact them for updates to their medical and family histories. Data and biospecimens will be stored for potential future research projects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or CT confirmed diagnosis of pancreatic adenocarcinoma
* Subjects with abnormal imaging study (CT, MRI, MRCP, EUS)
* Control subjects with a clinical diagnosis of a pancreas, liver, or intestinal condition
* Control subject with acute pancreatitis
* Control subject with chronic pancreatitis
* Control subject with biliary obstruction
* Control subject with pancreatic cyst
* Member of a high risk family (≥ 1 close relative with pancreatic cancer)
* Healthy control (without any of the above conditions)

Exclusion Criteria:

* Under the age of 18 years
* Unable to give informed consent
* Inability to travel to Pittsburgh for in-person enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who are diagnosed with pancreatic cancer, who are undergoing a procedure to evaluate their pancreas, and who have a family history of pancreatic cancer are recruited during appointments at the University of Pittsburgh Medical Center (e.g. Pancreas Specialty Care Center, GI laboratory, Hereditary GI Program)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2004-01; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The data will be used in cohort association studies. Endpoints will depend on the number of patients in the study and the number of markers that are being evaluated. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall E Brand, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States